CLINICAL TRIAL: NCT00499707
Title: A Randomized, Double-blind Trial to Evaluate the Efficacy and Safety of Fixed Dose Rosiglitazone/Metformin Combination Therapy Compared to Both Rosiglitazone and Metformin Monotherapies in Drug Naive Type 2 Diabetes Mellitus Subjects
Brief Title: Efficacy and Safety Study of Rosiglitazone/Metformin Therapy vs Rosiglitazone and Metformin in Type 2 Diabetes Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 712753/007
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: HbA1c; Drug-naive; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosiglitazone maleate/metformin hydrochloride — rosiglitazone maleate/metformin hydrochloride

SUMMARY:
The purpose of this 32 week study is to demonstrate that fixed-dose combination treatment with rosiglitazone/metformin will safely and effectively control glycemia as first line oral therapy in subjects type 2 diabetes. The primary objective of the study is to demonstrate superiority of rosiglitazone/metformin compared to its rosiglitazone and metformin.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Clinical diagnosis of type 2 diabetes
* HbA1c >7.5% to 11%
* FPG <270mg/dL (15mmol)
* Current treatment with diet and/or exercise alone, or no more than 15 days of an anti-diabetic medication or insulin within 12 weeks of screening

Exclusion Criteria:

* Clinically significant renal or hepatic disease
* Presence of anemia
* Presence of unstable or severe angina, coronary insufficiency, or any congestive heart failure requiring therapy
* Systolic blood pressure >170mmHg or diastolic blood pressure >100mmHg, while on anti-hypertensive treatment
* Chronic disease requiring intermittent or chronic treatment with corticosteroids
* Any female lactating, pregnant, or planning to become pregnant
* History of hepatocellular reaction, severe edema or a medically serious fluid related event associated with any thiazolidinedione
* Presence of acute or chronic metabolic acidosis
* History of diabetic ketoacidosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2003-10-08; Primary Completion 2004-12-01 (Actual); Study Completion 2004-12-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin A1c (HbA1c) at week 32. | at 32 week

SECONDARY OUTCOMES:
Key Secondary Measures: Change in FPG HbA1c and FPG responders Change in insulin, C-peptide, free fatty acids, lipids, insulin sensitivity and beta cell function Adverse Events Vital Signs Weight 32 weeks | at 32 weeksInvalid value

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (92):
- United States (44):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Los Banos, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Mogadore, Ohio
  - GSK Investigational Site, Downingtown, Pennsylvania
  - GSK Investigational Site, Warminster, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Australia (9):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Caulfield, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
  - GSK Investigational Site, Perth, Western Australia
- Brazil (2):
  - GSK Investigational Site, Recife, Pernambuco
  - GSK Investigational Site, São Paulo
- Canada (25):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Courtice, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Renfrew, Ontario
  - GSK Investigational Site, Stoney Creek, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Plessisville, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Saint Insidore de Dorchester, Quebec
  - GSK Investigational Site, Saint-Marc-des-Carrieres, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Mexico (5):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Mexico City
- New Zealand (4):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Rotorua
  - GSK Investigational Site, Wellington
- South Korea (3):
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Uijeongbu-si

REFERENCES:
- [Result] Chou H., et. al.; Rosiglitazone and metformin fixed-dose combination provides superior glycaemic control compared to metformin and rosiglitazone monotherapies, and was well tolerated in drug-naïve patients with T2DM [poster]; European Association for the Study of Diabetes, 10-15 September 2005, Athens, Greece.
- Available data/document: Informed Consent Form: 712753/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 712753/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 712753/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 712753/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 712753/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 712753/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 712753/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register